CLINICAL TRIAL: NCT01500187
Title: Fluoride Varnish Application for Treatment of White Spot Lesion After Fixed Orthodontic Treatment. A Pilot Study.
Brief Title: Fluoride Varnish for Treatment of White Spot Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Collaborators: University of Tennessee (Other); 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR-11-011; ORTHO2011-01 (Other: University of Tennessee)
Record Dates: First submitted 2011-12-22; First posted 2011-12-28 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: White Spot Lesions
Keywords: white spot lesions; fixed orthodontic brackets; fluoride varnish; fluoride gel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pediagel (Active Comparator): 1.23% Acidulated Phosphate Fluoride Gel
  Interventions: Device: Pediagel
- 3M Vanish Varnish (Experimental): 5% sodium fluoride varnish
  Interventions: Device: Vanish Varnish

INTERVENTIONS:
Device: Vanish Varnish — 5% sodium fluoride varnish with tricalcium phosphate
  Arms: 3M Vanish Varnish
Device: Pediagel — 1.23% Acidulated Phosphate Fluoride Gel
  Arms: Pediagel

SUMMARY:
Study will look at ability of fluoride varnish to remineralize white spot enamel lesions that can occur around the edge of fixed orthodontic brackets.

DETAILED DESCRIPTION:
To determine the efficacy of 5% sodium fluoride varnish with tricalcium phosphate in reverting white spot lesions after fixed orthodontic treatment, compared with a fluoride gel.

ELIGIBILITY:
Inclusion Criteria:

* no systemic disease
* has completed fixed orthodontic treatment, brackets debonded
* has at least two teeth with whitre spot lesions
* has received conventional periodontal therapy after orthodontic tretament

Exclusion Criteria:

* presence of enamel hypoplasia or dental fluorosis
* presence of tetracycline pigmentation
* periodontal pocketing of 3mm or greater
* taking antibiotics
* presence of carious cavities
* allergy to fluoride gel / varnish being used in study

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2012-02; Primary Completion 2014-03-31 (Actual); Study Completion 2014-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franklin Garcia-Godoy, DDS, MS, Principal Investigator — University of Tennessee
Locations (1):
- College of Dentistry, Memphis, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Teeth
Groups:
- Pediagel: 1.23% Acidulated Phosphate Fluoride Gel (Preventech)
- Vanish Varnish: 5% sodium fluoride varnish with tricalcium phosphate (3M)
Period: Overall Study
Arm/Group | Pediagel | Vanish Varnish
Started | 23; 106 Teeth | 15; 74 Teeth
Completed | 17; 76 Teeth | 15; 72 Teeth
Not Completed | 6; 30 Teeth | 0; 2 Teeth
Not completed — Lost to Follow-up | 6 | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: Teeth
Groups:
- Total: Total of all reporting groups
Arm/Group | Pediagel | Vanish Varnish | Total
Number analyzed (Participants) | 23 | 15 | 38
Number analyzed (Teeth) | 106 | 74 | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23 | 15 | 38
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 12 | 7 | 19

OUTCOME MEASURES:

1. Primary Outcome: DIAGNOdent Readings at Baseline, Three and Six Months - Intergroup Comparison
Description: Outcome of fluoride varnish or gel application to white spot lesions as measured by DIAGNOdent device after orthodontic debonding. Values shown represent the mean DIAGNOdent reading. The DIAGNOdent scale spans values from 0 to 30+ where larger values indicate higher levels of demineralization.
Time Frame: Baseline, Three and Six Month
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Teeth
Groups:
- Pediagel: 1.23% Acidulated phosphate fluoride
Arm/Group | Pediagel | Vanish Varnish
Number analyzed (Participants) | 15 | 15
Number analyzed (Teeth) | 76 | 72
units on a scale
  Baseline | 5.10 (2.67) | 6.01 (4.17)
  Three Months | 4.08 (2.32) | 5.50 (3.81)
  Six Months | 3.52 (2.46) | 3.95 (2.97)
Statistical Analysis 1: Comparison: Pediagel vs Vanish Varnish; Null Hypothesis: there is no intergroup difference (α=0.05) in DIAGNOdent reading at baseline; Test type: Superiority or Other; p = 0.636, ANOVA
Statistical Analysis 2: Comparison: Pediagel vs Vanish Varnish; Null Hypothesis: there is no intergroup difference (α=0.05) in DIAGNOdent reading at three months; Test type: Superiority or Other; p = 0.001, ANOVA
Statistical Analysis 3: Comparison: Pediagel vs Vanish Varnish; Null Hypothesis: there is no intergroup difference (α=0.05) in DIAGNOdent reading at six months; Test type: Superiority or Other; p = 0.423, ANOVA

ADVERSE EVENTS:
Time Frame: Six Months
Groups:
- Group 2: Oral B Minute-Gel, fluoride gel
  Oral B Minute-Gel: Fluoride gel
- Group 1: Vanish varnish, 5% sodium fluoride varnish with tricalcium phosphate
  Vanish varnish: 5% sodium fluoride varnish with tricalcium phosphate
Arm/Group | Group 2 | Group 1
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No